CLINICAL TRIAL: NCT01876706
Title: L.O.C.A.L. Study -- UroLift System TOlerability and ReCovery When Administering Local Anesthesia
Brief Title: UroLift System TOlerability and ReCovery When Administering Local Anesthesia
Acronym: LOCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeoTract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP12911
Record Dates: First submitted 2013-05-06; First posted 2013-06-13 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2019-03-20 (Actual); Status verified 2019-03

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: UroLift System
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UroLift® System (Experimental): Single-arm of qualified subjects receiving UroLift® System intervention.
  Interventions: Device: UroLift® System

INTERVENTIONS:
Device: UroLift® System — The NeoTract UroLift System is a medical device approved for sale in the European Union, Australia, and Canada. The UroLift® System is indicated for the treatment of symptoms due to urinary outflow obstruction secondary to benign prostatic hyperplasia (BPH) in men 50 years of age or older. During the procedure, an implant is delivered into the prostatic lobe obstructing the urethra and restricting urine flow. The distal end of the device is used to compress the lobe then the implant is delivered to retain the lobe in position, thereby increasing the urethral opening and reducing the fluid obstruction through the prostatic urethra.

SUMMARY:
The purpose of the study is to evaluate procedure tolerability and surgical recovery following the UroLift® system procedure when conducted with local anesthesia in subjects with symptomatic benign hyperplasia (BPH). Primary effectiveness will be achieved by looking at the Quality of Recovery Visual Analog Scale (QoR VAS) by the one month follow-up visit.

DETAILED DESCRIPTION:
The randomized portion of the study is a prospective, multicenter, non-blinded, single arm trial evaluating procedure tolerability and surgical recovery following the UroLift® system procedure when conducted with local anesthesia. All subjects undergo UroLift system treatment and will be followed through 5 years after receiving the investigational device.

ELIGIBILITY:
Inclusion Criteria:

* Males age of 50 years or older diagnosed with symptomatic benign prostatic hyperplasia (BPH)

Exclusion Criteria:

* Size, volume,length of prostate

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-04; Primary Completion 2014-10 (Actual); Study Completion 2018-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Shore, MD, Principal Investigator — Grand Strand Urology
Locations (7):
- United States (7):
  - Genesis Research LLC, San Diego, California
  - Advanced Urology Institute, Daytona Beach, Florida
  - Pinellas Urology, St. Petersburg, Florida
  - Chesapeake Urology, Baltimore, Maryland
  - Sheldon J. Freedman, M.D., Ltd., Las Vegas, Nevada
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Jean Brown Research, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- UroLift Arm: Subjects that undergo the UroLift System procedure
Period: Overall Study
Arm/Group | UroLift Arm
Started | 51
1 Month | 51
3 Months | 51
6 Months | 46
12 Months | 42
24 Months | 35
36 Months | 32
48 Months | 31
60 Months | 26
Completed | 26
Not Completed | 25
Not completed — BPH Intervention | 9
Not completed — Lost to Follow-up | 7
Not completed — Withdrawals | 6
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | UroLift Arm
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery
Description: Primary effectiveness will be achieved when 80% (95% lower confidence limit) of subjects achieve a score of 80 or more on the Quality of Recovery Visual Analog Scale (QoR VAS) by the one month follow-up visit. The VAS scale is 0-100, with 100 being 100% recovery.
Time Frame: 1 Month
Measure: Number; unit: participants
Arm/Group | UroLift Arm
Number analyzed (Participants) | 51
participants
  90 - 100 Score | 28
  80 - 89 Score | 16

2. Secondary Outcome: IPSS Scores at Baseline and 12 Month Follow-up
Description: The International Prostate Symptom Score (IPSS) is an 7 question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH). Lower scores are indicative of less symptoms.
  Score Correlation[1] 0-7 Mildly symptomatic 8-19 Moderately symptomatic 20-35 Severely symptomatic
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: IPSS total score
Arm/Group | UroLift Arm
Number analyzed (Participants) | 41
IPSS total score
  Baseline IPSS | 20.78 (5.28)
  12 Month IPSS | 9.73 (7.45)

3. Secondary Outcome: IPSS 12 Month Change From Baseline
Description: The International Prostate Symptom Score (IPSS) is an 7 question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH) using a total score from 0 - 35.
  The larger number for Change in IPSS Score 12 Month Follow-up from Baseline, demonstrate the improvement in IPSS.
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | UroLift Arm
Number analyzed (Participants) | 41
scores on a scale | 11.05 (7.15)

4. Secondary Outcome: IPSS 12 Month Percent (%) Change From Baseline
Description: The International Prostate Symptom Score (IPSS) is an 7 question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of the disease benign prostatic hyperplasia (BPH) using a total score from 0 - 35.
  The larger Percent (%) Change in IPSS Score at 12 Month Follow-up from Baseline, demonstrates the improvement in IPSS (the mean score was change by X %). Note: Percent (%) Change: is the mean % change of each subject.
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | UroLift Arm
Number analyzed (Participants) | 41
percentage change | 53.5 [43.1 to 63.9]

5. Secondary Outcome: BPH II Scores at Baseline and 12 Month Follow-up
Description: BPH Impact Index (BPH II) A validated questionnaire to measure how much urinary problems of patients with benign prostatic hyperplasia affect domains of health. BPHII total score is the combined (sum) of scores for Questions 1-4 (sum range of 0-13 scoring is presented below) MAX of 13 would be 3,3,3,and 4: A score of zero = Patient experiences no BPH impact and does not add any to score.
  Questions 1-4:
  1. Over the past month how much physical discomfort did any urinary problems cause you? &
  2. Over the past month, how much did you worry about your health because of any urinary problems? 0 None, 1, 2, 3 A lot.
  3. Overall, how bothersome has any trouble with urination been during the past month? 0 Not at all bothersome,1,2,3 Bothers me a lot.
  4. Over the past month, how much of the time has any urinary problems kept you from doing the kind of things you would usually do? 0 None of the time, 1,2,3, 4 All of the time.
Time Frame: 12 Month
Measure: Mean (Standard Deviation); unit: BPHII total score
Arm/Group | UroLift Arm
Number analyzed (Participants) | 41
BPHII total score
  Baseline BPHII | 6.32 (3.04)
  12 Month BPHII | 1.71 (2.30)

6. Secondary Outcome: BPH II 12 Month Percent (%) Change From Baseline
Description: as for outcome 5
Time Frame: 12 Months
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | UroLift Arm
Number analyzed (Participants) | 41
percentage change | 71.7 [61.2 to 82.2]

7. Secondary Outcome: BPH II 12 Month Change From Baseline
Description: as for outcome 5
Time Frame: 12 Months
Measure: Mean (Standard Deviation); unit: BPHII total score
Arm/Group | UroLift Arm
Number analyzed (Participants) | 41
BPHII total score | 4.61 (3.23)

8. Secondary Outcome: Qmax Scores at Baseline and 12 Month Follow-up
Description: QMAX indicates the maximum flow rate during a Uroflow in mL/sec. QMAX is used as an indicator for the diagnosis of enlarged prostate. A lower QMAX may indicate that the enlarged prostate puts pressure on the urethra.
Time Frame: 12 Month
Population: QMAX maximum peak urinary flow rate, if valid void >125ml at baseline and 12 months. Urinary flow rate overread by independent reviewer. Note that n=33 pertains to those subjects where a valid void was received, therefore 8 subject flows were either not valid or were not received.
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | UroLift Arm
Number analyzed (Participants) | 33
mL/sec
  Baseline Qmax | 8.33 (2.07)
  12 Month Qmax | 11.79 (4.50)

9. Secondary Outcome: QMAX 12 Month Change Minus Baseline
Description: QMAX indicates the maximum flow rate during a Uroflow in mL/sec. QMAX is used as an indicator for the diagnosis of enlarged prostate. A lower QMAX may indicate that the enlarged prostate puts pressure on the urethra. The larger number for Change of the QMAX value at 12 Month Follow-up minus Baseline, demonstrate the improvement in QMAX
Time Frame: 12 Months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mL/sec
Arm/Group | UroLift Arm
Number analyzed (Participants) | 33
mL/sec | 3.45 (4.58)

10. Secondary Outcome: QMAX 12 Month Percent (%) Change in mL/Sec From Baseline
Description: QMAX indicates the maximum flow rate during a Uroflow in mL/sec. QMAX is used as an indicator for the diagnosis of enlarged prostate. A lower QMAX may indicate that the enlarged prostate puts pressure on the urethra. The larger Percent (%) Change of the QMAX value at 12 Month Follow-up from Baseline, demonstrate the improvement in QMAX. Note: Percent (%) Change: is the average %change of each subject
Time Frame: 12 Months
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: percentage change
Arm/Group | UroLift Arm
Number analyzed (Participants) | 33
percentage change | 57.4 [17.9 to 97.0]

11. Secondary Outcome: Pain Tolerability Throughout the UroLift System Procedure
Description: Pain Tolerability using questionnaire pelvic pain Visual Analog Scale (VAS) 0-10. A score of 0 (zero) would equal no pain while a score of 10 would equate to pain as bad as patient could imagine. This scale was assessed at different times during procedure as specified in results section.
Time Frame: 12 Month
Population: Pain Tolerability throughout the UroLift System Procedure
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | UroLift Arm
Number analyzed (Participants) | 51
units on a scale
  During Flexible cystoscopy | 3.0 [0 to 10]
  After Rigid cystoscopy | 4.8 [0 to 10]
  During UroLift implant placement | 5.0 [0 to 10]
  After sheath removed (end of procedure) | 3.4 [0 to 10]

12. Secondary Outcome: BPHII Baseline and 12 Month Median Score, 95% CI
Description: as for outcome 5
Time Frame: 12 Month
Measure: Median (95% Confidence Interval); unit: BPHII total score
Arm/Group | UroLift Arm
Number analyzed (Participants) | 41
BPHII total score
  Baseline BPHII | 7.00 [5.36 to 7.28]
  12 Month BPHII | 1.00 [0.98 to 2.43]

13. Secondary Outcome: IPSS at Baseline and 12 Months, Median , 95% CI
Description: as for outcome 2
Time Frame: 12 Month
Measure: Median (95% Confidence Interval); unit: IPSS total score
Arm/Group | UroLift Arm
Number analyzed (Participants) | 41
IPSS total score
  Baseline IPSS score | 20.0 [19.11 to 22.45]
  12 Month IPSS score | 8.00 [7.38 to 12.08]

14. Secondary Outcome: QMAX Median at Baseline and 12 Months With CI 95%
Description: QMAX indicates the maximum flow rate during a Uroflow in mL/sec. QMAX is used as an indicator for the diagnosis of enlarged prostate. A lower QMAX may indicate that the enlarged prostate is obstructive.
Time Frame: 12 Month
Measure: Median (95% Confidence Interval); unit: mL/sec
Arm/Group | UroLift Arm
Number analyzed (Participants) | 33
mL/sec
  Baseline | 9.00 [7.60 to 9.07]
  12 Month | 12.0 [10.19 to 13.38]

ADVERSE EVENTS:
Time Frame: 5 Years;
Description: AEs reported from Index Procedure through 5 Year follow-up; No UADEs; No device or related SAEs
Arm/Group | UroLift Arm
All-Cause Mortality (participants affected / at risk) | 3/51
Serious Adverse Events (participants affected / at risk) | 12/51
Other Adverse Events (participants affected / at risk) | 47/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift Arm (N=51)
Congestive heart failure (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Lung mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Myocardial infarction (Cardiac disorders) | 2 (3)
Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastatic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Gallbladder necrosis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | UroLift Arm (N=51)
Hematuria (Renal and urinary disorders) | 42 (44)
Dysuria (Renal and urinary disorders) | 37 (46)
Pelvic pain (Reproductive system and breast disorders) | 12 (12)
Urge Incontinence (Renal and urinary disorders) | 15 (18)
Urinary urgency (Renal and urinary disorders) | 4 (6)
Urinary retention (Renal and urinary disorders) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (4)
Urinary frequency (Renal and urinary disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No